CLINICAL TRIAL: NCT04224428
Title: Role of Fexofenadine in Reducing Albuminurea in Patients With Diabetic Kidney Disease
Brief Title: Role of Fexofenadine in Diabetic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Basma Mahrous El-Fatatry, Principal investigator, Assistant lecturer of Clinical Pharmacy Department, Faculty of Pharmacy, Tanta University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FEXT20
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet
- Fexofenadine group (Active Comparator)
  Interventions: Drug: Fexofenadine Pill

INTERVENTIONS:
Drug: Fexofenadine Pill — fexofenadine tablets 60 mg once daily will be taken for six months
  Arms: Fexofenadine group
Drug: Placebo oral tablet — lactose oral tablet
  Arms: Control group

SUMMARY:
* This study will that will be conducted on 60 outpatients previously diagnosed with type 2 diabetes mellitus.
* Patients will be recruited from Internal Medicine Department, Tanta University Hospital, Tanta, Egypt.

This study will be randomized, controlled, parallel, prospective clinical study. Accepted patients will be randomized into 2 groups as the following

* Group 1 (Control group): 30 patients will receive maximum tolerated dose of ACEI for six months
* Group 2 (Fexofenadine group): 30 patients will receive maximum tolerated dose of ACEI plus fexofenadine tablets 60 mg once daily for six months

The primary end point will be the change in Urinary albumin to creatinine ratio (UACR) after six months of treatment

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥ 18 years
* Confirmed diagnosis of Type 2 diabetes mellitus at least 6 months prior to screening
* Stage 2 and 3 diabetic nephropathy (persistent micro- or macroalbuminuria with urinary albumin creatinine ratio (UACR) >30mg/g) despite treatment with maximum tolerated dose of ACE inhibitors for at least 8 weeks prior to the screening
* Hemoglobin A1c > 6.5 % with regular use of insulin and/or oral glucose lowering agents

Exclusion Criteria:

* Type 1 diabetes mellitus
* Severe renal impairment (eGFR< 30 mL/min/1.73 m2 at screening)
* Pregnant or lactating women
* Chronic heart failure
* Malignancy
* Inflammatory or autoimmune disease
* History of kidney disease other than diabetic nephropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Percent change in urinary albumin creatinine ratio (UACR) | After 6 months

SECONDARY OUTCOMES:
Urinary cyclophilin A | After 6 months
Urinary monocyte chemoattractant protein-1 (MCP-1) | After 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Fatatry BM, El-Haggar SM, Ibrahim OM, Shalaby KH. Repurposing fexofenadine as a promising candidate for diabetic kidney disease: randomized clinical trial. Int Urol Nephrol. 2024 Apr;56(4):1395-1402. doi: 10.1007/s11255-023-03804-w. Epub 2023 Sep 23. PMID 37741921